CLINICAL TRIAL: NCT06860061
Title: Changes of Corneal and Total Ocular Higher-Order Aberrations After Conventional LASIK, Femto-LASIK and PRK in Low and Moderate Myopia
Brief Title: Changes of Higher-Order Aberrations After Different Types of LASIK in Myopia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Abdeen Refai, Master degree ophthalmology department faculty of medicine Sohag University, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Soh-Med-24-12-4MD
Record Dates: First submitted 2025-02-19; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Conventional LASIK, Femto-LASIK and PRK in Low and Moderate Myopia

STUDY DESIGN:
Intervention Model Description: This prospective comparative interventional study will enroll patients with low and moderate myopia who seek laser vision correction at Sohag Center for LASIK and Corneal Surgeries, Sohag, Egypt. Eyes included will be divided into 3 groups according to the type of refractive surgery used (conventional LASIK, Femto-LASIK and PRK) and each group will be subdivided into 2 groups according to the degree of myopia (low and moderate).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1 (Active Comparator): Conventional Lasik
  Interventions: Procedure: Laser refractive surgery
- group 2 (Active Comparator): Femto LASIK
  Interventions: Procedure: Laser refractive surgery
- group 3 (Active Comparator): PRK
  Interventions: Procedure: Laser refractive surgery

INTERVENTIONS:
Procedure: Laser refractive surgery — This prospective comparative interventional study will enroll patients with low and moderate myopia who seek laser vision correction at Sohag Center for LASIK and Corneal Surgeries, Sohag, Egypt. Eyes included will be divided into 3 groups according to the type of refractive surgery used (conventional LASIK, Femto-LASIK and PRK) and each group will be subdivided into 2 groups according to the degree of myopia (low and moderate).
  All patients will be subjected to routine comprehensive preoperative examinations including manifest uncorrected distant visual acuity (UCDVA), best corrected distant visual acuity (BCDVA), slit-lamp examination, intraocular pressure, and fundus examination.
  Corneal topography and corneal aberrometry will be performed on all patients using Sirius's Scheimpflug-Placido topography (CSO, Florence, Italy). The CSO topography system analyzes a total of 6144 corneal points of a corneal area within a circular annulus outlined by an inner radius of 0.33 mm and an outer

SUMMARY:
This prospective comparative interventional study will enroll patients with low and moderate myopia who seek laser vision correction at Sohag Center for LASIK and Corneal Surgeries, Sohag, Egypt. Eyes included will be divided into 3 groups according to the type of refractive surgery used (conventional LASIK, Femto-LASIK and PRK) and each group will be subdivided into 2 groups according to the degree of myopia (low and moderate).

ELIGIBILITY:
Inclusion Criteria:

Age: 18 - 45 years old.

Refraction:

Low and moderate grades of myopia will be included:

(According to manifest refraction) low ([0] - ≤ [-3] diopters) Moderate ([-3] - ≤ [-6] diopters) With cylinder ≤ [-1.5] diopters.

Exclusion Criteria:

Any ocular surgery or medication, corneal opacities, pregnancy, lactation and keratoconus.

Ages: 18 Weeks to 45 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Changes of corneal higher-order aberrations | 1 year
  Corneal aberrometry will be performed using Sirius's Scheimpflug-Placido topography (CSO, Florence, Italy).
Changes of total ocular higher-order aberrations | 1 year
  Wavefront refraction will be acquired by the iDesign aberrometer (Hartmann-Shack Aberrometer)

IPD SHARING:
Plan to Share IPD: Undecided